CLINICAL TRIAL: NCT03872427
Title: A Phase II Basket Trial of Glutaminase Inhibitor (BEGIN) Telaglenastat (CB-839) HCL in Patients With NF1 Aberrations, NF1 Mutant Malignant Peripheral Nerve Sheath Tumors (MPNST), KEAP1/NRF2 and LKB1 Aberrant Tumors
Brief Title: Testing Whether Cancers With Specific Mutations Respond Better to Glutaminase Inhibitor, Telaglenastat Hydrochloride, Anti-Cancer Treatment, BeGIN Study
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NCI-2019-01365; NCI-2019-01365 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); NCI10220; 10220 (Other: University of Texas MD Anderson Cancer Center LAO); 10220 (Other: CTEP); UM1CA186688 (NIH)
Record Dates: First submitted 2019-03-12; First posted 2019-03-13 (Actual); Results first posted 2025-07-01 (Actual); Last update posted 2025-11-14 (Actual); Status verified 2025-10

CONDITIONS: Advanced Malignant Solid Neoplasm; Metastatic Malignant Solid Neoplasm; NF1 Mutation Positive Malignant Peripheral Nerve Sheath Tumor; Unresectable Malignant Solid Neoplasm
MeSH Terms: conditions — Neoplasm Metastasis | interventions — Specimen Handling; Magnetic Resonance Spectroscopy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Treatment (telaglenastat hydrochloride) (Experimental): Patients receive telaglenastat hydrochloride PO BID on days 1-28. Cycles repeat every 28 days in the absence of disease progression or unacceptable toxicity. Patients also undergo CT, MRI, or PET/CT during screening and on study, and collection of blood samples during screening and on study.
  Interventions: Procedure: Biospecimen Collection; Procedure: Computed Tomography; Procedure: Magnetic Resonance Imaging; Other: Pharmacodynamic Study; Procedure: Positron Emission Tomography; Drug: Telaglenastat Hydrochloride

INTERVENTIONS:
Procedure: Biospecimen Collection — Undergo collection of blood
  Other Names: Biological Sample Collection; Biospecimen Collected; Specimen Collection
Procedure: Computed Tomography — Undergo CT or PET/CT
  Other Names: CAT; CAT Scan; Computed Axial Tomography; Computerized Axial Tomography; Computerized axial tomography (procedure); Computerized Tomography; Computerized Tomography (CT) scan; CT; CT Scan; Diagnostic CAT Scan; Diagnostic CAT Scan Service Type; tomography
Procedure: Magnetic Resonance Imaging — Undergo MRI
  Other Names: Magnetic Resonance; Magnetic Resonance Imaging (MRI); Magnetic resonance imaging (procedure); Magnetic Resonance Imaging Scan; Medical Imaging, Magnetic Resonance / Nuclear Magnetic Resonance; MR; MR Imaging; MRI; MRI Scan; MRIs; NMR Imaging; NMRI; Nuclear Magnetic Resonance Imaging; sMRI; Structural MRI
Other: Pharmacodynamic Study — Correlative studies
  Other Names: PHARMACODYNAMIC; Pharmacodynamic (PD) study
Procedure: Positron Emission Tomography — Undergo PET/CT
  Other Names: Medical Imaging, Positron Emission Tomography; PET; PET Scan; Positron emission tomography (procedure); Positron Emission Tomography Scan; Positron-Emission Tomography; PT
Drug: Telaglenastat Hydrochloride — Given PO
  Other Names: CB-839 HCl; Glutaminase Inhibitor CB-839 Hydrochloride

SUMMARY:
This phase II trial studies how well glutaminase inhibitor telaglenastat hydrochloride (CB-839 HCl) works in treating patients with specific genetic mutations and solid tumors or malignant peripheral nerve sheath tumors that have spread to other places in the body (metastatic) or cannot be removed by surgery (unresectable). Glutaminase converts an amino acid (building block of proteins) called glutamine to glutamate, which can support several cellular pathways. Telaglenastat hydrochloride works by blocking glutamine activity needed for the growth of cells. When this activity is blocked, the growth of cancer cells may stop and the cancer cells may then die. Cancer is caused by changes (mutations) to genes that control the way cells function and uncontrolled cell growth may result in tumor formation. Specific genetic mutations studied in this clinical trial are NF1 mutation for malignant peripheral nerve sheath tumors, and NF1, KEAP1/NRF2, or STK11/LKB1 mutation for other solid tumors. Telaglenastat hydrochloride may stop the growth of tumor cells by blocking some of the enzymes needed for cell growth.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVE:

I. To assess the best overall response rate (BORR) achieved by 6 months of telaglenastat (CB-839) hydrochloride (HCl) treatment in specific pathway aberrant tumors (MPNST, NF1, KEAP1/NRF2 & STK11/ LKB1).

SECONDARY OBJECTIVES:

I. To determine the safety, progression-free survival (PFS), time to progression (TTP) and overall survival (OS).

II. To determine the overall response rate (ORR) (highest objective response achieved between start of therapy and progression), time to response (TTR) and clinical benefit rate (CBR) of telaglenastat (CB-839)HCl.

III. To assess pharmacodynamic changes and adaptive responses and correlate with response to treatment as well as disease progression (correlative objective).

EXPLORATORY OBJECTIVES:

I. Correlate fludeoxyglucose F-18 (18-F FDG) positron emission tomography (PET)/computed tomography (CT) pre-therapy and 8-weeks post-therapy response to telaglenastat (CB-839) HCl therapy.

II. Evaluate changes in level of circulating tumor deoxyribonucleic acid (DNA) at baseline, one month on-treatment and time of progression (Molecular Characterization Laboratory [MoCHA Labs]) to treatment response.

III. Quantify the peripheral blood concentrations of the metabolites: aspartate, glutamate, glutamine and arginine (@Mayo clinic Oncometabolomics core) and correlate with response.

IV. Evaluate the pharmacodynamic (PD) effect of telaglenastat (CB-839) HCl on systemic levels of the tricarboxylic acid (TCA) cycle metabolites in peripheral blood (baseline and one month) as part of the protocol.

V. Evaluate tumor by reverse phase protein array (@core facility at MD Anderson) and ribonucleic acid (RNA) sequencing (seq) to evaluate changes from pre-treatment, during treatment and post treatment specimens.

VI. Perform patient-derived tumor xenograft (PDX) modelling-co-clinical trials (@Dr. Funda Meric-Bernstam's lab MD Anderson) to understand response/resistance mechanisms and also evaluate combination therapies for future development.

OUTLINE:

Patients receive telaglenastat hydrochloride orally (PO) twice daily (BID) on days 1-28. Cycles repeat every 28 days in the absence of disease progression or unacceptable toxicity. Patients also undergo CT, magnetic resonance imaging (MRI), or PET/CT during screening and on study, and collection of blood samples during screening and on study.

After completion of study treatment, patients are followed up every 3 months thereafter.

ELIGIBILITY:
Inclusion Criteria:

* Patients must have histologically confirmed malignancy that is metastatic or unresectable
* Patient must have histopathologic confirmation of advanced solid tumor with NF1 mutation, NF1 mutant MPNST, KEAP1/NRF2 mutant and STK11/LKB1 mutant tumors (molecular profiling performed in any Clinical Laboratory Improvement Act [CLIA] certified lab [including tumor and circulating cell-free (cf)DNA], e.g. Caris, FoundationOne, FoundationAct, Oncomine, Guardant etc.)

  * NOTE: For all cohorts annotation for actionability will be performed by the PRECISION ONCOLOGY DECISION SUPPORT (PODS) TEAM SHEIKH KHALIFA BIN ZAYED AL NAHYAN INSTITUTE FOR PERSONALIZED CANCER THERAPY (IPCT) THE UNIVERSITY OF TEXAS MD ANDERSON CANCER CENTER 6565 MD ANDERSON BLVD, HOUSTON, TX 77030
* Patient must have no standard therapies available
* Patient must be aged greater than 18 years old for all cohorts
* Patients for NF1 mutant MPNST and NF1 mutant non-MPNST cohorts must be >= 40 kg
* Patient must be at least 4 weeks since any prior surgery or radiotherapy
* Females of childbearing potential must have a negative serum pregnancy test (=< 14 days) prior to start of trial treatment
* Response Evaluation Criteria in Solid Tumors (RECIST) measurable disease and biopsiable targetable lesion
* Patients must have measurable disease, defined as at least one lesion that can be accurately measured in at least one dimension (longest diameter to be recorded for non-nodal lesions and short axis for nodal lesions) as >= 20 mm (>= 2 cm) by chest x-ray or as >= 10 mm (>= 1 cm) with CT scan, magnetic resonance imaging (MRI), or calipers by clinical exam
* Patients with treated brain metastases are eligible if there is no evidence of progression for at least 4 weeks after central nervous system (CNS)-directed treatment, as ascertained by clinical examination and brain imaging (MRI or CT) during the screening period
* Human immunodeficiency virus (HIV)-infected patients on effective anti-retroviral therapy with undetectable viral load within 6 months are eligible for this trial
* Eastern Cooperative Oncology Group (ECOG) performance status =< 2 (Karnofsky >= 60%)
* Leukocytes >= 3,000/mcL
* Absolute neutrophil count >= 1,000/mcL
* Platelets >= 100,000/mcL
* Total bilirubin =< 1.5 x institutional upper limit of normal (ULN) and up to 3 ml/dL for patients with Gilbert's disease
* Aspartate aminotransferase (AST) (serum glutamic oxaloacetic transaminase [SGOT])/alanine aminotransferase (ALT) (serum glutamate pyruvate transaminase [SGPT]) =< 3 x institutional ULN and =< 5 x institutional ULN for patients with liver metastases
* Creatinine =< institutional ULN, as age appropriate OR
* Glomerular filtration rate (GFR) >= 30 mL/min/1.73 m^2 for patients with creatinine levels above institutional normal
* The effects of telaglenastat (CB-839) HCl on the developing human fetus are unknown. For this reason and because anti-metabolic agents like telaglenastat (CB-839) HCl are known to be teratogenic, women of child-bearing potential and men must agree to use adequate contraception (hormonal or barrier method of birth control; abstinence) prior to study entry and for the duration of study participation. Should a woman become pregnant or suspect she is pregnant while she or her partner is participating in this study, she should inform her treating physician immediately. Men treated or enrolled on this protocol must also agree to use adequate contraception prior to the study, for the duration of study participation, and 4 months after completion of telaglenastat (CB-839) HCl administration
* Ability to understand and the willingness to sign a written informed consent document

Exclusion Criteria:

* Patients who have had chemotherapy or radiotherapy within 4 weeks (6 weeks for nitrosoureas or mitomycin C) prior to entering the study
* Patients who have not recovered from adverse events due to prior anti-cancer therapy (i.e., have residual toxicities > grade 1)
* Patients who are receiving any other investigational agents
* History of allergic reactions attributed to compounds of similar chemical or biologic composition to telaglenastat (CB-839) HCl
* Patients with glioma will be excluded
* Patients with active or prior history of hepatitis B or C will be excluded
* Telaglenastat (CB-839) HCl is a weak in vitro inhibitor of CYP2C9. Therefore, patients receiving any medications or substances that are substrates of CYP2C9 are eligible, but should use caution with substrates that have a narrow therapeutic index. Because the lists of these agents are constantly changing, it is important to regularly consult a frequently-updated medical reference. As part of the enrollment/informed consent procedures, the patient will be counseled on the risk of interactions with other agents, and what to do if new medications need to be prescribed or if the patient is considering a new over-the-counter medicine or herbal product
* Uncontrolled intercurrent illness including, but not limited to, ongoing or active infection, symptomatic congestive heart failure, unstable angina pectoris, cardiac arrhythmia, or psychiatric illness/social situations that would limit compliance with study requirements
* Pregnant women are excluded from this study because telaglenastat (CB-839) HCl is anti-metabolic agent with the potential for teratogenic or abortifacient effects. Because there is an unknown but potential risk for adverse events in nursing infants secondary to treatment of the mother with telaglenastat (CB-839) HCl, breastfeeding should be discontinued if the mother is treated with telaglenastat (CB-839) HCl

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 54 (Actual)
Dates: Start 2019-12-14 (Actual); Primary Completion 2023-10-30 (Actual); Study Completion 2026-04-16 (Estimated)

CONTACTS AND LOCATIONS:
Overall Officials: Funda Meric-Bernstam, Principal Investigator — University of Texas MD Anderson Cancer Center LAO
Locations (31):
- United States (31):
  - University of Alabama at Birmingham Cancer Center, Birmingham, Alabama
  - UM Sylvester Comprehensive Cancer Center at Aventura, Aventura, Florida
  - UM Sylvester Comprehensive Cancer Center at Coral Gables, Coral Gables, Florida
  - UM Sylvester Comprehensive Cancer Center at Deerfield Beach, Deerfield Beach, Florida
  - University of Miami Miller School of Medicine-Sylvester Cancer Center, Miami, Florida
  - UM Sylvester Comprehensive Cancer Center at Kendall, Miami, Florida
  - UM Sylvester Comprehensive Cancer Center at Plantation, Plantation, Florida
  - Moffitt Cancer Center-International Plaza, Tampa, Florida
  - Moffitt Cancer Center - McKinley Campus, Tampa, Florida
  - Moffitt Cancer Center, Tampa, Florida
  - Northwestern University, Chicago, Illinois
  - University of Kansas Clinical Research Center, Fairway, Kansas
  - HaysMed, Hays, Kansas
  - University of Kansas Cancer Center, Kansas City, Kansas
  - The University of Kansas Cancer Center - Olathe, Olathe, Kansas
  - Mercy Hospital Pittsburg, Pittsburg, Kansas
  - Salina Regional Health Center, Salina, Kansas
  - University of Kansas Health System Saint Francis Campus, Topeka, Kansas
  - University of Kansas Hospital-Westwood Cancer Center, Westwood, Kansas
  - University of Kentucky/Markey Cancer Center, Lexington, Kentucky
  - National Cancer Institute Developmental Therapeutics Clinic, Bethesda, Maryland
  - National Institutes of Health Clinical Center, Bethesda, Maryland
  - Dana-Farber Cancer Institute, Boston, Massachusetts
  - University Health Truman Medical Center, Kansas City, Missouri
  - Laura and Isaac Perlmutter Cancer Center at NYU Langone, New York, New York
  - NYP/Columbia University Medical Center/Herbert Irving Comprehensive Cancer Center, New York, New York
  - Wake Forest University at Clemmons, Clemmons, North Carolina
  - Wake Forest University Health Sciences, Winston-Salem, North Carolina
  - Ohio State University Comprehensive Cancer Center, Columbus, Ohio
  - University of Pittsburgh Cancer Institute (UPCI), Pittsburgh, Pennsylvania
  - M D Anderson Cancer Center, Houston, Texas

IPD SHARING:
Plan to Share IPD: Yes
NCI is committed to sharing data in accordance with NIH policy. For more details on how clinical trial data is shared, access the link to the NIH data sharing policy page
URL: https://grants.nih.gov/policy/sharing.htm

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Out of the 55 patients enrolled, one patient did not receive treatment due to a death before starting the trial.
Groups:
- Cohort 1: NF1 mutant malignant peripheral nerve sheath tumors (MPNST)
- Cohort 2: NF1 mutant other cancers
- Cohort 3: KEAP1/NRF2 mutant cancers
- Cohort 4: STK11/LKB1 mutant cancers
Period: Overall Study
Arm/Group | Cohort 1 | Cohort 2 | Cohort 3 | Cohort 4
Started | 9 | 26 | 9 | 10
Completed | 9 | 26 | 9 | 10
Not Completed | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Cohort 1 | Cohort 2 | Cohort 3 | Cohort 4 | Total
Number analyzed (Participants) | 9 | 26 | 9 | 10 | 54
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0 | 0
  Between 18 and 65 years | 7 | 12 | 7 | 8 | 34
  >=65 years | 2 | 14 | 2 | 2 | 20
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 4 | 17 | 4 | 5 | 30
  Male | 5 | 9 | 5 | 5 | 24
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1 | 0 | 0 | 1 | 2
  Not Hispanic or Latino | 8 | 26 | 9 | 9 | 52
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0
  Asian | 0 | 0 | 1 | 1 | 2
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0
  Black or African American | 5 | 2 | 1 | 1 | 9
  White | 4 | 24 | 7 | 7 | 42
  More than one race | 0 | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0 | 1 | 1
Region of Enrollment [Number; unit: participants]
  United States | 9 | 26 | 9 | 10 | 54

OUTCOME MEASURES:

1. Primary Outcome: Best Overall Response Rate by 6 Months
Description: Best overall response rate (BORR) based on RECIST V1.1 achieved by 6 months of CB-839 HCl treatment
Time Frame: Up to 6 months from treatment start date
Measure: Count of Participants; unit: Participants
Arm/Group | Cohort 1 | Cohort 2 | Cohort 3 | Cohort 4
Number analyzed (Participants) | 9 | 26 | 9 | 10
Participants
  Complete Response (CR)/Partial response (PR) | 0 | 1 | 0 | 0
  Stable Disease (SD) | 4 | 10 | 2 | 4
  Progressive disease (PD) | 4 | 14 | 6 | 5
  Treatment Failure | 1 | 1 | 1 | 1

2. Secondary Outcome: Incidence of Adverse Events
Description: Will be assessed by Common Terminology Criteria for Adverse Events version 5.0. Will tabulate toxicity by cohort, type, severity and attribution.
Time Frame: Up to 2 years from treatment start date
Reporting Status: Not Posted

3. Secondary Outcome: Progression-free Survival
Description: Will estimate using the Kaplan-Meier method with time zero set to cycle 1, day 1 (C1D1). Will estimate the medians and select probabilities along with 95% confidence intervals. If more than a handful of patients die without progression, will use Aalen-Johansen estimates to adjust for the competing risk of death.
Time Frame: Time to progression or death whichever comes first, assessed up to 2 years from treatment start date
Reporting Status: Not Posted

4. Secondary Outcome: Time to Progression
Description: Will estimate the medians and select probabilities along with 95% confidence intervals. If more than a handful of patients die without progression, will use Aalen-Johansen estimates to adjust for the competing risk of death.
Time Frame: Time to progression starting at C1D1, assessed up to 2 years from treatment start date
Reporting Status: Not Posted

5. Secondary Outcome: Overall Survival
Description: Will estimate using the Kaplan-Meier method with time zero set to C1D1. Will estimate the medians and select probabilities along with 95% confidence intervals. If more than a handful of patients die without progression, will use Aalen-Johansen estimates to adjust for the competing risk of death.
Time Frame: Time to death from any cause, assessed up to 2 years from treatment start date
Reporting Status: Not Posted

6. Secondary Outcome: Overall Response Rate
Time Frame: From start of treatment until disease progression/recurrence, assessed up to 2 years
Reporting Status: Not Posted

7. Secondary Outcome: Clinical Benefit Rate
Time Frame: Up to 2 years from treatment start date
Reporting Status: Not Posted

8. Other Pre Specified Outcome: Pharmacodynamic (PD) Tumor Oncometabolite Levels of Glutamine
Description: Will assess PD changes before and after treatment using the Wilcoxon signed rank test. Will correlate these changes with response to treatment using Wilcoxon rank sum test. Will also perform a receiver operating characteristic curve analysis.
Time Frame: Baseline up to between 0-8 hours post-glutaminase inhibitor CB-839 hydrochloride dose
Reporting Status: Not Posted

9. Other Pre Specified Outcome: PD Tumor Oncometabolite Levels of Glutamate
Description: as for outcome 8
Time Frame: Baseline up to between 0-8 hours post-glutaminase inhibitor CB-839 hydrochloride dose
Reporting Status: Not Posted

10. Other Pre Specified Outcome: PD Tumor Oncometabolite Levels of Aspartate
Description: as for outcome 8
Time Frame: Baseline up to between 0-8 hours post-glutaminase inhibitor CB-839 hydrochloride dose
Reporting Status: Not Posted

ADVERSE EVENTS:
Time Frame: 4 years
Arm/Group | Cohort 1 | Cohort 2 | Cohort 3 | Cohort 4
All-Cause Mortality (participants affected / at risk) | 7/9 | 20/26 | 6/9 | 8/10
Serious Adverse Events (participants affected / at risk) | 5/9 | 7/26 | 4/9 | 6/10
Other Adverse Events (participants affected / at risk) | 9/9 | 24/26 | 8/9 | 10/10
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Cohort 1 (N=9) | Cohort 2 (N=26) | Cohort 3 (N=9) | Cohort 4 (N=10)
Abdominal pain (Gastrointestinal disorders) | 0 | 1 | 1 | 0
Acute kidney injury (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0
Appendicitis (Gastrointestinal disorders) | 0 | 1 | 0 | 0
Ascites (Gastrointestinal disorders) | 0 | 1 | 0 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0
Bacteremia (Blood and lymphatic system disorders) | 0 | 1 | 0 | 0
Blood bilirubin increased (Blood and lymphatic system disorders) | 0 | 1 | 0 | 0
Chest wall pain (Cardiac disorders) | 1 | 0 | 0 | 0
Colonic obstruction (Gastrointestinal disorders) | 0 | 0 | 1 | 0
Constipation (Gastrointestinal disorders) | 0 | 0 | 2 | 2
Death NOS (General disorders) | 1 | 2 | 0 | 2
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 2
Encephalopathy (Nervous system disorders) | 0 | 1 | 0 | 0
Esophageal obstruction (Gastrointestinal disorders) | 0 | 0 | 0 | 1
Fever (General disorders) | 0 | 1 | 0 | 0
Gait disturbance (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1
General and admin site - Other - Failure To Thrive (General disorders) | 0 | 1 | 0 | 1
Generalized edema (General disorders) | 0 | 0 | 0 | 1
Generalized muscle weakness (General disorders) | 0 | 1 | 0 | 0
Hypercalcemia (Blood and lymphatic system disorders) | 0 | 1 | 0 | 0
Hypoglycemia (Metabolism and nutrition disorders) | 1 | 0 | 0 | 0
Hyponatremia (Blood and lymphatic system disorders) | 0 | 0 | 1 | 0
Hypoxia (General disorders) | 0 | 0 | 1 | 0
Lung infection (Infections and infestations) | 0 | 1 | 0 | 0
Nausea (Gastrointestinal disorders) | 1 | 0 | 0 | 0
Nervous system - Other - L5 Lumbar Lesion Compress Nerve Route (Nervous system disorders) | 1 | 0 | 0 | 0
Non-cardiac chest pain (General disorders) | 1 | 0 | 0 | 0
Pain (General disorders) | 0 | 2 | 1 | 0
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 1
Resp, thoracic & mediast - Other - Hemoptysis (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0
Tracheal obstruction (Gastrointestinal disorders) | 2 | 0 | 0 | 0
Tumor pain (General disorders) | 0 | 1 | 1 | 0
Vomiting (Gastrointestinal disorders) | 1 | 0 | 0 | 0
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Cohort 1 (N=9) | Cohort 2 (N=26) | Cohort 3 (N=9) | Cohort 4 (N=10)
ALT increased (Investigations) | 2 | 11 | 1 | 0
Abdominal pain (Gastrointestinal disorders) | 1 | 6 | 1 | 2
Alkaline phosphatase increased (Investigations) | 1 | 8 | 0 | 1
Anemia (Blood and lymphatic system disorders) | 2 | 10 | 5 | 3
Anorexia (Metabolism and nutrition disorders) | 2 | 5 | 3 | 3
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 | 2 | 0 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 1 | 2 | 0 | 2
Bladder infection (Infections and infestations) | 1 | 0 | 0 | 0
Bruising (General disorders) | 1 | 0 | 0 | 1
Chest wall pain (Cardiac disorders) | 1 | 0 | 0 | 0
Chills (General disorders) | 1 | 1 | 0 | 0
Cholesterol high (Investigations) | 1 | 0 | 0 | 0
Concentration impairment (Nervous system disorders) | 1 | 0 | 0 | 0
Constipation (Gastrointestinal disorders) | 2 | 6 | 2 | 2
Cough (Respiratory, thoracic and mediastinal disorders) | 3 | 1 | 0 | 1
Creatinine increased (Investigations) | 1 | 4 | 1 | 1
Dehydration (Metabolism and nutrition disorders) | 1 | 2 | 0 | 2
Diarrhea (Gastrointestinal disorders) | 1 | 2 | 0 | 1
Dizziness (Nervous system disorders) | 1 | 1 | 0 | 0
Dysgeusia (Gastrointestinal disorders) | 1 | 0 | 1 | 0
Dysphagia (Gastrointestinal disorders) | 1 | 1 | 0 | 0
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 3 | 2 | 1 | 3
Ear and Labyrinth - Other - Decreased Hearing (Ear and labyrinth disorders) | 1 | 0 | 0 | 0
Edema face (General disorders) | 1 | 0 | 0 | 0
Eye disorders - Other, specify - Sty (Eye disorders) | 1 | 0 | 0 | 0
Fall (General disorders) | 2 | 1 | 0 | 1
Fatigue (General disorders) | 5 | 9 | 1 | 3
Fever (General disorders) | 1 | 2 | 0 | 0
General and admin site - Other - Migraine (General disorders) | 1 | 0 | 0 | 0
General and admin site - Other - Sleep Disorder (General disorders) | 1 | 0 | 0 | 0
Headache (Nervous system disorders) | 2 | 3 | 1 | 1
Hypercalcemia (Metabolism and nutrition disorders) | 1 | 5 | 3 | 0
Hyperglycemia (Metabolism and nutrition disorders) | 1 | 2 | 1 | 2
Hyperkalemia (Metabolism and nutrition disorders) | 2 | 2 | 0 | 1
Hypertension (Vascular disorders) | 1 | 2 | 0 | 1
Hypoalbuminemia (Metabolism and nutrition disorders) | 1 | 1 | 2 | 1
Hypoglycemia (Metabolism and nutrition disorders) | 1 | 0 | 0 | 0
Hyponatremia (Metabolism and nutrition disorders) | 5 | 7 | 4 | 4
Hypophosphatemia (Metabolism and nutrition disorders) | 2 | 1 | 2 | 0
Infections & infestations - Other - Covid (Infections and infestations) | 1 | 0 | 0 | 0
Infections & infestations - Other - Covid-19 (Infections and infestations) | 1 | 0 | 0 | 0
Injury/poison/procedure - Other - Dislocation Of Rib (Left) (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0
Insomnia (Psychiatric disorders) | 2 | 2 | 1 | 0
Irregular menstruation (Reproductive system and breast disorders) | 1 | 0 | 0 | 0
Lymphocyte count decreased (Investigations) | 4 | 10 | 2 | 3
Memory impairment (Nervous system disorders) | 1 | 1 | 0 | 0
Metabolism and nutrition - Other - Positive For Appetite Change (Metabolism and nutrition disorders) | 1 | 0 | 0 | 0
Muscle cramp (Musculoskeletal and connective tissue disorders) | 1 | 1 | 0 | 0
Musculoskel/connect tissue -Other - Right Hip Pain (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0
Musculoskel/connect tissue -Other - Shaking At Night (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0
Musculoskel/connect tissue -Other - Tumor Pain (Back) (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0
Myalgia (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0
Nausea (Gastrointestinal disorders) | 3 | 9 | 1 | 3
Neck pain (Musculoskeletal and connective tissue disorders) | 1 | 1 | 0 | 0
Neutrophil count decreased (Investigations) | 2 | 5 | 0 | 0
Non-cardiac chest pain (General disorders) | 1 | 2 | 0 | 1
Pain (General disorders) | 2 | 2 | 1 | 1
Peripheral motor neuropathy (Nervous system disorders) | 1 | 2 | 0 | 1
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0
Reproductive and breast - Other - Abnormal Image Finding (Reproductive system and breast disorders) | 1 | 0 | 0 | 0
Reproductive and breast - Other - Sclerosing Intraductal Papilloma Without Atypia (Reproductive system and breast disorders) | 1 | 0 | 0 | 0
Skin & subcutaneous tissue -Other - Cellulitis (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0
Skin & subcutaneous tissue -Other - Joint Swelling (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0
Skin & subcutaneous tissue -Other - Skin Infection (Cut/Right Foot Wound) (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0
Skin papilloma (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0
Trismus (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0
Tumor pain (General disorders) | 1 | 1 | 0 | 0
Voice alteration (General disorders) | 1 | 0 | 0 | 0
Vomiting (Gastrointestinal disorders) | 2 | 6 | 0 | 1
Weight gain (Metabolism and nutrition disorders) | 1 | 0 | 0 | 0
Weight loss (Metabolism and nutrition disorders) | 2 | 4 | 3 | 1
White blood cell decreased (Investigations) | 2 | 5 | 0 | 1
AST increased (Investigations) | 0 | 8 | 1 | 1
Abdominal distension (Gastrointestinal disorders) | 0 | 1 | 0 | 1
Activated PTT prolonged (Investigations) | 0 | 1 | 0 | 0
Allergic reaction (General disorders) | 0 | 1 | 0 | 0
Bacteremia (Blood and lymphatic system disorders) | 0 | 1 | 0 | 0
Blood bilirubin increased (Blood and lymphatic system disorders) | 0 | 3 | 0 | 0
Blood/Lymph - Other - Neutropenia (Blood and lymphatic system disorders) | 0 | 1 | 0 | 0
Bronchial infection (Infections and infestations) | 0 | 1 | 0 | 0
Cholecystitis (Gastrointestinal disorders) | 0 | 1 | 0 | 0
Depression (Psychiatric disorders) | 0 | 1 | 0 | 0
Dry eye (Eye disorders) | 0 | 1 | 0 | 0
Dry mouth (Gastrointestinal disorders) | 0 | 1 | 0 | 0
Dry skin (Skin and subcutaneous tissue disorders) | 0 | 1 | 1 | 1
Ear and Labyrinth - Other - Hyperacusis (Ear and labyrinth disorders) | 0 | 1 | 0 | 0
Edema limbs (General disorders) | 0 | 1 | 1 | 0
Elevated LDH (Investigations) | 0 | 4 | 2 | 0
Eye disorders - Other, specify - Visual Disturbance (Eye disorders) | 0 | 1 | 0 | 0
Floaters (Eye disorders) | 0 | 2 | 0 | 0
GI disorders - Other, specify - Heartburn (Gastrointestinal disorders) | 0 | 1 | 0 | 0
Gastroesophageal reflux disease (Gastrointestinal disorders) | 0 | 1 | 0 | 0
Generalized muscle weakness (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0
Hiccups (Gastrointestinal disorders) | 0 | 1 | 0 | 0
Hypocalcemia (Metabolism and nutrition disorders) | 0 | 1 | 0 | 0
Hypokalemia (Metabolism and nutrition disorders) | 0 | 1 | 0 | 1
Hypomagnesemia (Metabolism and nutrition disorders) | 0 | 2 | 0 | 0
Hypotension (Vascular disorders) | 0 | 1 | 0 | 0
Infections & infestations - Other - Covid19 Positive (Infections and infestations) | 0 | 1 | 0 | 0
Lipase increased (Investigations) | 0 | 1 | 0 | 0
Malaise (General disorders) | 0 | 1 | 0 | 1
Metabolism and nutrition - Other - Lactic Acidosis (Metabolism and nutrition disorders) | 0 | 1 | 0 | 0
Metabolism and nutrition - Other - Metabolic Acidosis (Metabolism and nutrition disorders) | 0 | 1 | 0 | 0
Mucositis oral (Gastrointestinal disorders) | 0 | 1 | 0 | 0
Nervous system - Other - Numbness To Bilateral Foot R>L (Nervous system disorders) | 0 | 1 | 0 | 0
Neuralgia (Nervous system disorders) | 0 | 1 | 0 | 0
Oral dysesthesia (Gastrointestinal disorders) | 0 | 1 | 0 | 0
Pain in extremity (General disorders) | 0 | 2 | 0 | 1
Paresthesia (Nervous system disorders) | 0 | 1 | 0 | 0
Periorbital edema (General disorders) | 0 | 1 | 0 | 0
Photophobia (Nervous system disorders) | 0 | 6 | 1 | 0
Platelet count decreased (Investigations) | 0 | 5 | 2 | 2
Pruritus (Skin and subcutaneous tissue disorders) | 0 | 1 | 1 | 0
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 0
Rhinorrhea (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0
Serum amylase increased (Investigations) | 0 | 1 | 0 | 0
Shingles (Infections and infestations) | 0 | 1 | 0 | 0
Sinus tachycardia (Cardiac disorders) | 0 | 1 | 1 | 0
Skin & subcutaneous tissue -Other - Itching (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 0
Stomach pain (Gastrointestinal disorders) | 0 | 1 | 0 | 0
Toothache (Gastrointestinal disorders) | 0 | 1 | 0 | 0
Tremor (General disorders) | 0 | 1 | 0 | 0
Urinary frequency (Renal and urinary disorders) | 0 | 1 | 0 | 0
Urinary tract infection (Infections and infestations) | 0 | 1 | 0 | 0
Bone pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0
Confusion (Nervous system disorders) | 0 | 0 | 1 | 0
INR increased (Investigations) | 0 | 0 | 1 | 0
Muscle weakness lower limb (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0
Rectal pain (Gastrointestinal disorders) | 0 | 0 | 1 | 0
Renal & urinary disorders - Other - Difficulty Urination (Renal and urinary disorders) | 0 | 0 | 1 | 0
Wheezing (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 1
Adrenal insufficiency (General disorders) | 0 | 0 | 0 | 1
Anxiety (Psychiatric disorders) | 0 | 0 | 0 | 1
Delirium (Nervous system disorders) | 0 | 0 | 0 | 1
Hoarseness (General disorders) | 0 | 0 | 0 | 1
Hypoxia (General disorders) | 0 | 0 | 0 | 1
Investigations - Other, specify - Ldh Increase (Investigations) | 0 | 0 | 0 | 1
Localized edema (General disorders) | 0 | 0 | 0 | 1
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1
Rash acneiform (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 1
Resp, thoracic & mediast - Other - Hypoxemia (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1
Resp, thoracic & mediast - Other - Pulmonary Opacities (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1
Seroma (General disorders) | 0 | 0 | 0 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2025-01-03): https://cdn.clinicaltrials.gov/large-docs/27/NCT03872427/Prot_SAP_001.pdf
  • Informed Consent Form (2025-01-03): https://cdn.clinicaltrials.gov/large-docs/27/NCT03872427/ICF_002.pdf